CLINICAL TRIAL: NCT06421870
Title: Renoprotective Effects of Dapagliflozin Versus Pentoxiphylline in Chronic Kidney Disease Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, nahla mohamed elsayed teama, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD277/2023
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Dapagliflozin; Chronic kidney disease; Pentoxiphylline
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin; Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin arm (Active Comparator): 70 patients will take dapagliflozin 10 mg per day for 1 year in addition to standard management for chronic kidney disease
  Interventions: Drug: Dapagliflozin 10mg Tab
- Pentoxiphylline arm (Active Comparator): 70 patients will take pentoxifylline 400 mg twice daily for 1 year in addition to standard management for chronic kidney disease
  Interventions: Drug: Pentoxifylline 400 MG
- Control (No Intervention): 70 patients won't take either dapagliflozin or pentoxiphylline but they will continue their standard management for chronic kidney disease

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Patients will be given dapagliflozin 10 mg once daily
  Arms: Dapagliflozin arm
Drug: Pentoxifylline 400 MG — Patients will be given pentoxyifylline 400 mg twice daily
  Arms: Pentoxiphylline arm

SUMMARY:
Kidneys have a vital role in glucose homeostasis by various mechanisms, one of the major mechanisms is through SGLT2. This role was commonly overlooked till development of the new SGLT2 inhibitors. (Ni, L., et al 2020) The SGLT2 inhibitor class of glucose-lowering agents has recently shown beneficial effects to reduce the onset and progression of renal complications in people with and without diabetes, through slow the decline in glomerular filtration rate (GFR), delaying the onset of microalbuminuria and slow or reverse the progression of proteinuria. (Nespoux, J., & Vallon, V. 2020) The drug pentoxifylline is a methyl-xanthine derivative and a nonselective phosphodiesterase inhibitor with anti-inflammatory, antiproliferative and antifibrotic actions currently indicated for peripheral artery disease. (Panchapakesan U et al.,2018) Chronic kidney disease is a progressive disorder in which patients are treated according to complications presented such as hypocalcemia, hyperkalemia, anemia and metabolic acidosis.

DETAILED DESCRIPTION:
It is only in recent years that the attention was drawn on the key role of the kidney in glucose homeostasis. Nevertheless, along with the liver, the kidney has a key role in ensuring the energy needs during fasting periods. This organ has a vital role in absorbing the entire quantity of the filtered glucose. Having a glomerular filtration rate of 180 litres per day, it filters approximately 180 grams of glucose per day, bringing its contribution in maintaining normal fasting plasma glucose (FPG) levels. (Cersosimo, E.et al 2014) The reabsorption of glucose is ensured by the sodium-glucose cotransporter (SGLT) 2, responsible for the reabsorption of 90% of glucose, and SGLT1, that reabsorbs the remaining glucose. (Mota, M., et al 2015) Glomerular hyperfiltration is a common pathway of kidney injury both in diabetic and non-diabetic settings and is associated with progression of kidney function decline. (Hoogeveen, E. K. 2022) Sodium-glucose co-transporter-2 (SGLT2) inhibitors are glucose-lowering agents that eliminate excess glucose through a glucosuric effect by reducing glucose reabsorption from the renal filtrate (Thomson, S. C., et al. 2019) It is indicated that the expression of high mobility group box 1 (HMGB1) increased in patients with kidney disease, and may result in renal injury through the activation of nuclear factor- κB (NF- κB) and an increase in receptor for advanced glycation end products (RAGE) expression. It is suggested that Dapagliflozin achieves its reno-protective status through its antioxidative stress and anti-inflammatory action via inhibition of the HMGB1 - RAGE - NF- κB signalling pathway. (Yao, D et al., 2018) SGLT2 is found almost exclusively in the luminal membranes of epithelial cells lining the first and second segments of the proximal tubules, where it mediates reabsorption of most (typically ≥ 90%) of filtered glucose. (Mudaliar S, et al. 2015) By inhibiting SGLT2 beneficial kidney effects are thought to be mediated by various mechanisms, including restoration of tubule-glomerular feedback leading to a reduction in intraglomerular pressure and hyperfiltration. Both conditions are considered core components of the pathophysiology contributing to progression of diabetic as well as nondiabetic CKD. Reductions in intraglomerular pressure, as shown by agents blocking the renin-angiotensin system, are frequently accompanied by a hemodynamic acute decrease in GFR, which is reversible after treatment cessation. (Wanner et al., 2018).

Common drug side effects of dapagliflozin include urinary tract infections, cystitis, hypotension, dehydration and female genital mycotic infections. Hypoglycemic episodes were reported in 6% to 10% of patients who administer dapagliflozin concurrently with insulin and insulin secretagogues. (Anderson SL et al., 2014) Pentoxifylline (PTF) is a synthetic dimethylxanthine derivative that modulates the rheological properties of blood and has both anti-oxidant and anti-inflammatory properties. PTF has been investigated for its possible use in diverse conditions, including osteoradionecrosis, diabetic kidney disease, and generally any condition associated with fibrosis. (Wen WX et al., 2017) PTF reduces levels of inflammatory markers: high-sensitivity C-reactive protein (hs-CRP), serum fibrinogen and TNF-α, this could reduce albuminuria and slow renal disease progression. (de Morales AM et al, 2019)

Thus, we need to evaluate the effect of Dapagliflozin versus Pentoxifylline on GFR among CKD non-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 2 and 3

Exclusion Criteria:

* Diabetes mellitus
* History of recurrent or recent genitourinary infections
* Immunosuppressive medications
* Malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate | 1 year
  eGFR will be based on serum creatinine and will be calculated by CKD-EPI 2021
Change in proteinuria | 1 year
  Proteinuria quantification done by urine protein to creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Saeed A Saeed, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Ni L, Yuan C, Chen G, Zhang C, Wu X. SGLT2i: beyond the glucose-lowering effect. Cardiovasc Diabetol. 2020 Jun 26;19(1):98. doi: 10.1186/s12933-020-01071-y. PMID 32590982
- [Background] Nespoux J, Vallon V. Renal effects of SGLT2 inhibitors: an update. Curr Opin Nephrol Hypertens. 2020 Mar;29(2):190-198. doi: 10.1097/MNH.0000000000000584. PMID 31815757
- [Background] Panchapakesan U, Pollock C. Drug repurposing in kidney disease. Kidney Int. 2018 Jul;94(1):40-48. doi: 10.1016/j.kint.2017.12.026. Epub 2018 Apr 6. PMID 29628139
- [Background] Cersosimo E, Solis-Herrera C, Triplitt C. Inhibition of renal glucose reabsorption as a novel treatment for diabetes patients. J Bras Nefrol. 2014 Jan-Mar;36(1):80-92. doi: 10.5935/0101-2800.20140014. PMID 24676619
- [Background] DeFronzo RA, Davidson JA, Del Prato S. The role of the kidneys in glucose homeostasis: a new path towards normalizing glycaemia. Diabetes Obes Metab. 2012 Jan;14(1):5-14. doi: 10.1111/j.1463-1326.2011.01511.x. PMID 21955459